CLINICAL TRIAL: NCT05544903
Title: The Use of Point of Care Ultrasound to Predict Intensive Care Unit Admission of Patients Presenting With Sepsis to the Emergency Department
Brief Title: Point of Care Ultrasound to Predict Intensive Care Unit Admission of Patients Presenting With Sepsis to the Emergency Department
Acronym: POCUS Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Northwell Health (Other)
Collaborators: Flosonics Medical (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20-0151
Record Dates: First submitted 2022-09-09; First posted 2022-09-19 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mortality, ICU admission, or rapid response team activation: Carotid flow patterns and velocity time integral values, as determined by FloPatch.
- No mortality, ICU admission, or rapid response team activation: Carotid flow patterns and velocity time integral values, as determined by FloPatch.

SUMMARY:
The FloPatch device will be applied to 150 septic patients in the emergency department before they receive fluid resuscitation. This study will assess whether initial FloPatch measured volume-responsiveness and volume of fluids used will predict a composite outcome of mortality, intensive care unit admission, or rapid response team activation. The development of fluid unresponsiveness throughout the initial fluid resuscitation will be assessed and its association with the composite outcome will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department patient
* 18+ years old
* Systolic blood pressure less than 100mmHg
* Respiratory rate greater than 22 breaths per minutes
* Temperature greater than 38 degrees Celsius or less than 36 degrees Celsius
* Heart rate greater than 90 beats per minute

Exclusion Criteria:

* Already intubated prior to emergency department arrival
* Ventilator-dependent
* Patients transferred from another hospital
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department who meet sepsis criteria based on presenting vital signs will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Mortality | 24 hours
  This study will ascertain whether the patient died within 24 hours of ED arrival.
ICU admission | 24 hours
  This study will ascertain whether the patient was admitted to the ICU within 24 hours of ED arrival.
Rapid response team activation | 24 hours
  This study will ascertain whether a rapid response team was activated for the patient within 24 hours of ED arrival.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Cohen, MD, Principal Investigator — North Shore University Hospital
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No